CLINICAL TRIAL: NCT01609621
Title: Tibiopedal Access for Crossing of Infrainguinal Artery Occlusions
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-008
Record Dates: First submitted 2012-05-16; First posted 2012-06-01 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Retrograde access
  Interventions: Device: Retrograde tibiopedal arterial access

INTERVENTIONS:
Device: Retrograde tibiopedal arterial access — Retrograde, percutaneous arterial access of vessels at or below the tibioperoneal trunk, using a 21 gage needle or micropuncture introducer set, to facilitate crossing and treatment (e.g., angioplasty, stenting, atherectomy) of occlusive arterial lesions in the lower limb.

SUMMARY:
The objective of this prospective, non-randomized, multicenter, post-market, observational study is to compile clinical data on percutaneous techniques used to obtain tibiopedal access and to cross infrainguinal arterial occlusions.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a totally occluded infrainguinal artery, due to peripheral arterial atherosclerotic disease, for which a previous attempt to cross the occlusion using an antegrade approach was unsuccessful. For institutions where tibiopedal access is performed as a primary standard-of-care procedure, a prior unsuccessful antegrade approach attempt is not required.

Exclusion Criteria:

* Patient will not sign the Informed Consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected among those presenting with symptoms of peripheral arterial ischemic disease of the lower extremities and for whom endovascular intervention is deemed appropriate.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Technical Success deeming tibial pedal arterial access | 1 - 4 hours post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Walker, MD, Principal Investigator — Terrebone General Medical Center
Locations (11):
- United States (8):
  - Interventional Technologies, LLC (Tucson Medical Center), Tucson, Arizona
  - MedStar Health Research Institute (Washington Hospital Center), Washington D.C., District of Columbia
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - University of Miami (Mount Sinai Hospital), Miami, Florida
  - Terrebone Medical Center, Houma, Louisiana
  - Metro Heart and Vascular, Wyoming, Michigan
  - Rex Hospital, Inc, Raleigh, North Carolina
  - CAMC Health Education and Research Institute, Inc., Charleston, West Virginia
- Germany (2):
  - Universit ts-Herzzentrum Freiburg - Bad Krozingen GmbH, Bad Krozingen
  - Park-Krankenhaus Leipzig GmbH, Leipzig
- Casa Di Cura Abano Terme, Abano Terme, Italy

REFERENCES:
- [Derived] Walker CM, Mustapha J, Zeller T, Schmidt A, Montero-Baker M, Nanjundappa A, Manzi M, Palena LM, Bernardo N, Khatib Y, Beasley R, Leon L, Saab FA, Shields AR, Adams GL. Tibiopedal Access for Crossing of Infrainguinal Artery Occlusions: A Prospective Multicenter Observational Study. J Endovasc Ther. 2016 Dec;23(6):839-846. doi: 10.1177/1526602816664768. Epub 2016 Aug 24. PMID 27558463